CLINICAL TRIAL: NCT02824367
Title: Evaluation of Clinical Perfectionism in Parkinson Disease
Acronym: EPMP-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2014_843_0002; 2013-A01302-43 (Other: ID-RCB)
Record Dates: First submitted 2014-04-22; First posted 2016-07-06 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Perfectionism
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parkinsonian (Other): Patient Arm: Parkinsonian will complete several scale of evaluation. Behavioral: Completion of scales evaluation
  Interventions: Behavioral: Completion of scales evaluation
- Dystonic (Other): Comparator Arm: Dystonic patient will complete several scale of evaluation. Behavioral: Completion of scales evaluation
  Interventions: Behavioral: Completion of scales evaluation

INTERVENTIONS:
Behavioral: Completion of scales evaluation — Patient complete scores to perfectionism scales (Frost Multidimensional Perfectionism Scales (FMPS), Hewitt Multidimensional Perfectionism Scale (HMPS), scores to depression scale (Beck Depression Inventory (BDI)) and anxiety scale (State Trait Anxiety Inventory (STAI))

SUMMARY:
Scientific studies show that almost half of the people with Parkinson's Disease (PD) suffer of depression and / or anxiety.

DETAILED DESCRIPTION:
Scientific studies show that almost half of the people with Parkinson's Disease (PD) suffer of depression and / or anxiety. Also, clinicians reported that they exhibit specific personality traits (e.g., rigidity and perfectionism).

To date, few studies used Cognitive Behavioural Therapies (CBT) in people with Parkinson's disease showing promising results. Recently, perfectionism has received particular attention because of it association with many emotional disorders. Thus, some psychometric tools have been developed in order to evaluate different aspects of perfectionism. Yet, none of them has been used in people with Parkinson's disease.

The objective of this study is to investigate whether there is a direct link between Parkinson's disease and perfectionism by using psychometric tools from the CBT literature. Identifying such link would allow to justify the use of CBT in people with Parkinson's disease with the goal in mind to improve their care and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Score Mini Mental Scale (MMS) greater than 23
* For Parkinsonian, Parkinson disease be defined according to the criteria of the Unified Parkinson Disease Rating Scale (UPDRS), with a Hoehn and Yahr stage 1, 2 or 3
* The control patients present dystonias not within the scope of Parkinson
* Informed Consent Form signed
* Patient covered by social insurance

Exclusion Criteria:

* Proven Presence of neuropsychological disorders
* Patients with deep brain stimulation
* Diagnosis of somatic pathology diagnosed
* Private Patient freedom or protected adult (under guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Perfectionism evaluation 1 | Day 0
  Scores to perfectionism scales (Frost Multidimensional Perfectionism Scales (FMPS)
Perfectionism evaluation 2 | Day 0
  Hewitt Multidimensional Perfectionism Scale (HMPS).

SECONDARY OUTCOMES:
Depression and anxiety evaluation 1 | Day 0
  Scores to depression scale (Beck Depression Inventory (BDI))
Depression and anxiety evaluation 2 | Day 0
  anxiety scale (State Trait Anxiety Inventory (STAI))

CONTACTS AND LOCATIONS:
Overall Officials: Pierre KRYSTKOWIAK, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France